CLINICAL TRIAL: NCT01119885
Title: Fentanyl Matrix for the Treatment of Pain Caused by Osteoarthritis of the Knee or Hip: Improvement of Pain and Function: Multicenter, Open-label, Prospective, Observational Study
Brief Title: Observational Study Investigating the Effectiveness of Fentanyl Matrix in Relieving Pain and Improving Function in Patients With Osteoarthritis of the Knee or Hip
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015454
Record Dates: First submitted 2010-01-29; First posted 2010-05-10 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Pain; Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: chronic pain; fentanyl matrix; arthritis; osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis, Hip; Osteoarthritis, Knee; Chronic Pain; Arthritis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 001: fentanyl matrix Knee osteoarthritis starting with 12mcg/h (flexible dose)
  Interventions: Drug: fentanyl matrix
- 002: fentanyl matrix Hip osteoarthritis starting with 12mcg/h (flexible dose)
  Interventions: Drug: fentanyl matrix

INTERVENTIONS:
Drug: fentanyl matrix — Knee osteoarthritis, starting with 12mcg/h (flexible dose)
  Groups: 001
Drug: fentanyl matrix — Hip osteoarthritis, starting with 12mcg/h (flexible dose)
  Groups: 002

SUMMARY:
The purpose of this study is to investigate the utility of fentanyl matrix for the treatment of pain due to osteoarthritis (OA) of knee or hip, which was not adequately controlled by non-opioid analgesic (e.g. NSAIDs or COX-II inhibitors) or weak opioids [tramadol HClacetaminophen, tramadol or codeine (or combinations with acetaminophen/ibuprofen)].

DETAILED DESCRIPTION:
This study is a prospective, open-label, non-interventional study. The objective of this study is to investigate the utility of fentanyl matrix after 8 week treatment of fentanyl matrix for the treatment of pain due to osteoarthritis (OA) of knee or hip, which was not adequately controlled by non-opioid analgesic (e.g. NSAIDs or COX-II selective inhibitors) or weak opioids [tramadol HCl with acetaminophen, tramadol or codeine (or combination with acetaminophen/ibuprofen)] in clinical practice according to the investigator's discretion. This study will investigate the usefulness of fentanyl matrix based on improvement in pain and function after Fentanyl matrix administration in patients who complained of pain caused by osteoarthritis and indicated for Fentanyl matrix administration in clinical practice at the investigator's discretion. This study will also measure the patients' functional improvement through Korean Version of WOMAC. Observational study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients who complain of chronic pain caused by osteoarthritis of the knee or hip persisting for 3 months or longer
* Patients who can fully observe the overall clinical study requirements including K-WOMAC completion at the investigator's discretion
* Patients who complain of severe pain (NRS score = 7) because pain was not treated enough with the previous analgesic
* Patients who have never been administered strong opioid analgesics over the last one month

Exclusion Criteria:

* Patients with a history of the drug or alcohol abuse in the past or now
* Childbearing women who are pregnant or likely to be pregnant during the study period and male subjects who are neither infertile nor willing to refrain from sexual relations but whose partner does not conduct an effective contraception (implant, injections, oral contraceptives, intrauterine device, etc.)
* Patients who are unable to use a transdermal system due to skin disease
* Patients with serious mental disorder
* Patients with history of hypersensitivity to opioid analgesics
* Patients with history of CO2 retention
* Patients who are not eligible for the study participation based on warnings, precautions and contra medications in the package insert of the study drug at the investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is the patients who visit a center during the study period with the complaint of chronic pain caused by osteoarthritis of the knee or hip, and are deemed to fail to control pain in a proper way and need fentanyl matrix administration according to the investigator's discretion
Sampling Method: Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity from baseline through final evaluation as measured by Numeric Rating Scale | Baseline and week 8

SECONDARY OUTCOMES:
Improved pain relief as measured using the K-WOMAC scale | baseline, week 4 and week 8
Improvement of sleep disturbance | baseline, week 4 and week 8
Impact of activity of daily activities measured by 5-point likert scale and social activities measured by 5-point likert scale | baseline, week 4 and week 8
Investigator and patient global assessment measured by 5-point likert scale | Week 4 and week 8
Improved pain relief as measured using the CGI-I | Week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.